CLINICAL TRIAL: NCT03548857
Title: Muscle Function After Lung Transplantation in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Acronym: COPD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Camilla Koch Ryrsø, Principle Investigator, Rigshospitalet, Denmark
Other Study IDs: H-17039327
Record Dates: First submitted 2018-05-09; First posted 2018-06-07 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: COPD
Keywords: Muscle dysfunction; Cardiovascular regulation; Lung transplantation (LTx)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Lung Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples (plasma), muscle biopsies (m. quadriceps femoris), transbronchial biopsy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COPD patients: COPD patients on the waiting list for a lung transplantation
  Interventions: Other: Lung transplantation

INTERVENTIONS:
Other: Lung transplantation — Single or double lung transplantation in patients with COPD

SUMMARY:
The purpose of the project is to investigate changes in the quadriceps muscle and cardiovascular regulation during exercise in relation to improved lung function after lung transplantation in patients with COPD.

DETAILED DESCRIPTION:
Dysfunctional skeletal musculature of the lower limbs is related to low quality of life, exercise intolerance and higher mortality in patients with COPD. Limb muscle dysfunction in COPD consists of muscle atrophy and reduced muscle strength but also intra-muscular alterations in oxidative capacity and mitochondrial function are often present. Moreover, reduced blood flow to exercising muscle may also contribute to the muscle dysfunction in COPD. The mechanisms responsible for muscle dysfunction in COPD patients remain unclear but could be a consequence of reduced lung function, inflammation, medications or low physical activity. Loss of lung function with COPD is normally irreversible so the transition to near-normal lung function after lung transplantation is a unique model to investigate the adaptation of the limb muscle to improved lung function. Thus, the purpose of this project is to investigate the effect of lung transplantation on limb muscle function (mitochondrial function, oxidative enzyme capacity, fiber type distribution, oxygen delivery/uptake) and daily physical activity level in patients with COPD. The project has a translational focus on muscle dysfunction in COPD and uses methodologies from clinical medicine, integrative physiology and molecular biochemistry in order to gain knowledge of mechanisms behind limb muscle dysfunction and exercise intolerance in COPD.

ELIGIBILITY:
Inclusion Criteria:

* COPD with or without alpha 1-antitrypsin deficiency on the waiting list for a lung transplantation
* Single or double lung transplantation
* ≥ 18 years
* Ability to give informed consent

Exclusion Criteria:

* Retransplantation
* Multiple-organ transplantation (heart-lung transplantation)
* Musculoskeletal disorders which substantially inhibits physical activity
* Need for crossmatching in connection with lung transplantation
* Anticoagulant therapy before lung transplantation (except acetylsalicylic acid)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: COPD patients on the waiting list for a lung transplantation
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-08-20 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in leg blood flow (mL/min) | Change from baseline at 6 months
  Endothelium function will be evaluated during acute exercise (one legged kicking) by Flow doppler
Change in 6 min walking test | Change from baseline at 6 months
  Exercise capacity
Change in health-related quality of life | Change from baseline at 6 months
  Health-related quality of life will be assessed by total mean score of St. George's Respiratory Questionnaire (SGRQ) (2 parts,3 components questionnaire). Scores range from 0 to 100, with higher scores indicating more limitations. A minimum change in score of 4 units are considered clinically relevant.
Change in health-related quality of life | Change from baseline at 6 months
  Health-related quality of life will be assessed by mean score of a validated Danish version of the COPD Assessment Test (CAT). The CAT is a short 8-item questionnaire with scoring range of 0-40, where higher scores indicating more limitations. A change of 2 units suggests a meaningful difference.

SECONDARY OUTCOMES:
Change in skeletal muscle function | Change from baseline at 6 months
  Muscle biopsy
Change in blood volume | Change from baseline at 6 months
  CO re-breathing method
Change in capillarization of lung tissue | Change from baseline at 6 months
  Transbronchial biopsy (only COPD patients)

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik Winning Iepsen, MD, PhD, Principal Investigator — Centre for Physical Activity Research, Copenhagen University Hospital, Copenhagen, Denmark
Locations (1):
- the Centre for Physical Activity Research, Copenhagen University Hospital, Copenhagen, Denmark